CLINICAL TRIAL: NCT01739985
Title: Postoperative Vomiting in Children: Evaluation of the Addition of Droperidol to Conventional Bi-prophylaxis
Brief Title: Postoperative Vomiting in Children: Comparison Tri - Versus bi -Prophylaxis
Acronym: VPOP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P081228; 2009-017293-20 (EudraCT Number)
Record Dates: First submitted 2012-07-20; First posted 2012-12-04 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2013-08

CONDITIONS: Postoperative Vomiting
Keywords: Postoperative; Vomiting; Children; Prophylaxis; Droperidol; Ondansetron; Dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Dexamethasone; Ondansetron; Droperidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone + ondansetron + Placebo (Active Comparator): dexamethasone + ondansetron + Placebo
  Interventions: Drug: Dexamethasone + ondansetron + Placebo
- Dexamethasone + ondansetron + Droperidol (Experimental): dexamethasone + ondansetron + Droperidol
  Interventions: Drug: Dexamethasone + ondansetron + Droperidol

INTERVENTIONS:
Drug: Dexamethasone + ondansetron + Placebo — Administration of ondansetron and dexamethasone immediately after induction of anesthesia. Ondansetron is administered at a dose of 100 micrograms.kg-1, dexamethasone at a dose of 125 microg x kg-1.Administration of the saline 30 minutes before the end of surgery
  Arms: Dexamethasone + ondansetron + Placebo
Drug: Dexamethasone + ondansetron + Droperidol — Administration of ondansetron and dexamethasone immediately after induction of anesthesia. Ondansetron is administered at a dose of 100 micrograms.kg-1, dexamethasone at a dose of 125 microg x kg-1Administration of droperidol 30 minutes before surgery at a dose of 50 micrograms.kg-1
  Arms: Dexamethasone + ondansetron + Droperidol

SUMMARY:
The purpose of this study is to evaluate the benefit of addition of droperidol to prophylaxis with ondansetron and dexamethasone in children with high risk of postoperative vomiting (POV). In adults some authors showed that the effectiveness of prophylaxis is correlated to the number of molecules or specific procedures used.

DETAILED DESCRIPTION:
The overall incidence of postoperative vomiting between 25 and 30% for the pediatric population, but it can reach a much higher incidence associated with certain types of surgery, about 80% in some studies like strabismus surgery for example. The identification of patients at high risk of POV is possible through the use of risk score. It is currently only one pediatric validated risk score, but the investigators conducted a multicenter study on this subject, whose results are being analyzed. This should allow us to identify children at high risk of POV. In this targeted population, the prophylaxis should allow a significant reduction in the incidence of POV. In children only one study tried to evaluate the association of ondansetron, dexamethasone and droperidol to prevent postoperative vomiting. However, different doses of the different molecules were combined, the extremely complicated design of this study and important methodological bias do not provide evidence about the superiority of the combination of three anti-emetics compared with two anti-emetics. Our present randomized, double-blind study is designed to compare the effectiveness of Droperidol in combination with a conventional bi-prophylaxis (dexamethasone/ondansetron) to the conventional bi-prophylaxis alone to decrease the occurrence of postoperative vomiting in children at high risk. The combination ondansetron and dexamethasone is frequently assessed as an association to prevent postoperative vomiting also in the adult population and in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for surgery and with high risk of postoperative vomiting, i.e. with VPOP score up to 4
* Between 3 to 18 years
* Informed consent signed or the owner (s) of parental
* Children receiving a social security system

Exclusion Criteria:

* Ambulatory surgery
* Preoperative corticosteroids
* Postoperative sedation
* Allergy known to droperidol, ondansetron or dexamethasone
* Known hypokaliemia
* Known hypomagnesemia
* Bradycardia (<55 bpm)
* Congenital long QT syndrome
* Treatment that induce prolonged QT
* Pheochromocytoma
* Severe depressive syndrome

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 322 (Actual)
Dates: Start 2010-12; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Postoperative vomiting | 24 hours

SECONDARY OUTCOMES:
Safety and Tolerability | 24 hours
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Gilles ORLIAGUET, MD, PhD, Study Chair — Necker Hospital
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Background] Gunter JB, McAuliffe JJ, Beckman EC, Wittkugel EP, Spaeth JP, Varughese AM. A factorial study of ondansetron, metoclopramide, and dexamethasone for emesis prophylaxis after adenotonsillectomy in children. Paediatr Anaesth. 2006 Nov;16(11):1153-65. doi: 10.1111/j.1460-9592.2006.01952.x. PMID 17040305
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Derived] Bourdaud N, Francois C, Jacqmarcq O, Guye ML, Jean J, Studer C, Engrand-Donal C, Devys JM, Boutin F, Guyot E, Bouazza N, Treluyer JM, Orliaguet GA; VPOP2 group. Addition of droperidol to prophylactic ondansetron and dexamethasone in children at high risk for postoperative vomiting. A randomized, controlled, double-blind study. Br J Anaesth. 2017 Jun 1;118(6):918-923. doi: 10.1093/bja/aex099. PMID 28505233